CLINICAL TRIAL: NCT03304314
Title: Assessment of Pupillary Response and Visual Field Defects by Objective Multifocal Chromatic Pupillometer in Patients With Pseudotumor Cerebri and Healthy Subjects
Brief Title: Multifocal Chromatic Pupilloperimetry in Patients With Pseudotumor Cerebri and Healthy Subjects.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Dr. Ygal Rotenstreich, Head of ElectrophisiologyClinic and Retinal Research Laboratory, Sheba Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: SHEBA-17-3754-YR-CTIL
Record Dates: First submitted 2017-09-17; First posted 2017-10-09 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Pseudotumor Cerebri
Keywords: PTC; EYES; Pseudotumor cerebri; increased Intracranial pressure; ICP
MeSH Terms: conditions — Pseudotumor Cerebri; Intracranial Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pseudotumor cerebri (PTC) patients (Experimental)
  Interventions: Diagnostic Test: objective chromatic multifocal pupillometer
- Control (Experimental)
  Interventions: Diagnostic Test: objective chromatic multifocal pupillometer

INTERVENTIONS:
Diagnostic Test: objective chromatic multifocal pupillometer — objective chromatic multifocal pupillometer (OCMP) enables objective and accurate measurement of pupillary responses to chromatic light at different wavelengths and light intensities and at different visual field locations.

SUMMARY:
PTC(Pseudotumor cerebri) patients may develop increased Intracranial pressure (ICP) that can produces increased pressure around the distal optic nerve,which is likely followed by venule compression, ischemia, and loss of visual function.Vision loss in PTC is most commonly characterized by standard automated perimetry to measure peripheral visual field sensitivity.

Pupillometry is a promising approach for functional assessment in PTC because it is noninvasive, objective, performed quickly with minimal patient cooperation needed.

The feasibility of using chromatic multifocal pupillometry for assesment of PTC will be examined.

ELIGIBILITY:
Inclusion Criteria:

Healthy subjects

1. Male or female patients, age between 18 and 80 years, inclusive
2. Informed written consent will be obtained from all participants.
3. Normal eye examination
4. Best-corrected visual acuity (BCVA) of 20/20
5. Normal color vision test (Ishihara/HRR)
6. Normal Spectral-Domain Optical Coherence Tomography (SD-OCT)
7. Normal 24-2 Humphrey visual field (SITA Standard) and:

   * Short duration (≤10 minutes)
   * Minimal fixation losses, False POS errors and False NEG errors (less than 33% for each one of reliability indices)

PTC patients

1. Male or female patients, age between 18 and 80 years, inclusive
2. Best-corrected visual acuity (BCVA) of at least 20/100 in worse eye
3. Optic disc edema
4. PTC diagnosis based on Modified Dandy Criteria ( lumbar puncture with opening pressure higher than or equal to 25 cm H2O, normal cerebrospinal fluid constituents, and unremarkable brain imaging results except typical for PTC

Exclusion Criteria:

Healthy subjects

1. History of past (last 3 months) or present ocular disease or ocular surgery
2. Use of any topical or systemic medications that could adversely influence pupillary reflex
3. Intolerance to gonioscopy, slit lamp examination, Goldmann applanation tonometry or other schedule study procedure.
4. Mental impairment or instability such as that informed consent may not be obtained or compliance with tester instructions is unlikely.
5. Visual media opacity including cloudy corneas.
6. Any condition preventing accurate measurement or examination of the pupil.

PTC patients

1. Any other neurologic or ophthalmic disease other than PTC
2. Use of any topical or systemic medications that could adversely influence pupillary reflex
3. Intolerance to gonioscopy, slit lamp examination, Goldmann applanation tonometry or other schedule study procedure.
4. Mental impairment or instability such as that informed consent may not be obtained or compliance with tester instructions is unlikely.
5. Visual media opacity including cloudy corneas.
6. Any condition preventing accurate measurement or examination of the pupil.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-11-03 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Measurement of maximal precentage of pupil contraction and dilation in response to chromatic light stimulus | single visit: 1 day
  Percentage of pupil contraction and dilation in response to blue and red light displayed at 76 test targets in a visual field of 30 degree will be measured in PTC patients and compared to matched controls
Measurement of maximal velocity of pupil contraction and dilation in response to chromatic light stimulus | single visit: 1 day
  Pupil contraction and dilation velocity (in pixel/second) in response to blue and red light displayed at 76 test targets in a visual field of 30 degree will be measured in PTC patients and compared to matched controls
Measurement of latency of pupil contraction and dilation in response to chromatic light stimulus | single visit: 1 day
  Pupil contraction and dilation latency (in seconds) in response to blue and red light displayed at 76 test targets in a visual field of 30 degree will be measured in PTC patients and compared to matched controls

SECONDARY OUTCOMES:
Subjective visual field | single visit: 1 day
  Humphrey perimetry
Optic nerve structure by OCT | single visit: 1 day
  OCT imaging
Change from baseline pupil contraction and dilation precentage in PCT patients at 48 hours | single visit: 1 day, 48 hours after baseline testing
  The change in percentage of pupil contraction and dilation in response to blue and red light displayed at 76 test targets in a visual field of 30 degree will be measured in PTC patients 48 hours after baseline measurement
Change from baseline pupil contraction and dilation maximal velocity in PCT patients at 48 hours | single visit: 1 day, 48 hours after baseline testing
  The change in maximal velocity of pupil contraction and dilation in response to blue and red light displayed at 76 test targets in a visual field of 30 degree will be measured in PTC patients 48 hours after baseline measurement
Change from baseline pupil contraction and dilation latency in PCT patients at 48 hours | single visit: 1 day, 48 hours after baseline testing
  The change in latency of pupil contraction and dilation in response to blue and red light displayed at 76 test targets in a visual field of 30 degree will be measured in PTC patients 48 hours after baseline measurement
Change from baseline pupil contraction and dilation precentage in PCT patients at 1 week. | single visit: 1 day, 1 week after baseline testing
  The change in percentage of pupil contraction and dilation in response to blue and red light displayed at 76 test targets in a visual field of 30 degree will be measured in PTC patients 1 weeks after baseline measurement
Change from baseline pupil contraction and dilation maximal velocity in PCT patients at 1 week. | single visit: 1 day, 1 week after baseline testing
  The change in maximal velocity of pupil contraction and dilation in response to blue and red light displayed at 76 test targets in a visual field of 30 degree will be measured in PTC patients 1 week after baseline measurement
Change from baseline pupil contraction and dilation latency in PCT patients at 1 week. | single visit: 1 day, 1 week after baseline testing
  The change in latency of pupil contraction and dilation in response to blue and red light displayed at 76 test targets in a visual field of 30 degree will be measured in PTC patients 1 week after baseline measurement
Change from baseline pupil contraction and dilation precentage in PCT patients at 2 months. | single visit: 1 day, 2 months after baseline testing
  The change in percentage of pupil contraction and dilation in response to blue and red light displayed at 76 test targets in a visual field of 30 degree will be measured in PTC patients 2 months after baseline measurement
Change from baseline pupil contraction and dilation maximal velocity in PCT patients at 2 months. | single visit: 1 day, 2 months after baseline testing
  The change in maximal velocity of pupil contraction and dilation in response to blue and red light displayed at 76 test targets in a visual field of 30 degree will be measured in PTC patients 2 months after baseline measurement
Change from baseline pupil contraction and dilation latency in PCT patients at 2 months. | single visit: 1 day, 2 months after baseline testing
  The change in latency of pupil contraction and dilation in response to blue and red light displayed at 76 test targets in a visual field of 30 degree will be measured in PTC patients 2 months after baseline measurement

CONTACTS AND LOCATIONS:
Locations (1):
- Sheba Medical Center, Tel Litwinsky, Israel

IPD SHARING:
Plan to Share IPD: No